CLINICAL TRIAL: NCT00919126
Title: An International Phase III Randomised Trial Comparing the Propofol Consumption During General Anaesthesia With Xenon in Inspiratory Concentrations of 50% and 70% and Total I.V. Anaesthesia Alone in ASA III Patients With Increased Risk of Perioperative Cardiac Complications.
Brief Title: General Anesthesia With Xenon in Inspiratory Concentrations of 50% and 70% and Total I.V. Anaesthesia.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment rate
Sponsor: Air Liquide SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALMED-07-C3-007; 2007-001979-10
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Anaesthesia
Keywords: Xenon in Anaesthesia
MeSH Terms: interventions — Xenon; Air; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Xenon 50% (45%-55%) in Oxygen (45%-55%),
  Interventions: Drug: Xenon
- Group B (Experimental): Xenon 70% (65%-75%) in Oxygen (25%-35%)
  Interventions: Drug: Xenon
- Group C (Active Comparator): Medical Air in Oxygen (45%-55%)
  Interventions: Drug: Medical Air in Oxygen

INTERVENTIONS:
Drug: Xenon — Maintenance of anaesthesia obtained with Xenon 50% and propofol infusion adjusted to depth of anaesthesia.
  Arms: Group A
Drug: Xenon — Maintenance of anaesthesia obtained with Xenon 70% and propofol infusion adjusted to depth of anaesthesia.
  Arms: Group B
Drug: Medical Air in Oxygen — Maintenance of anaesthesia obtained with propofol infusion adjusted to depth of anaesthesia.
  Arms: Group C

SUMMARY:
The purpose of this study is to evaluate the quantity of propofol administered with Xenon in two inspiratory concentrations, to maintain comparable depth of anaesthesia during the maintenance period of general anaesthesia.

DETAILED DESCRIPTION:
The inert or "noble" gas Xenon has anaesthetic properties that have been recognized 50 years ago. Several preclinical studies and investigations using xenon as an inhalational anaesthetic in humans were performed and reported that this gas has many properties of the ideal anaesthetic agent. Moreover, it is known that when xenon is combined with volatile anaesthetics or opioids, the required doses of those substances are reduced, resulting in a lower incidence of side effects. Patients could benefit from the administration of xenon if this inspired concentration would result in reduced doses of co-administered drugs.

This trial should allow evaluating the propofol consumption required in combination with xenon administered in inspiratory concentrations of 50% and 70% to maintain comparable depth of general anaesthesia as total i.v. anaesthesia, in ASA III patients presenting increased risk of perioperative cardiac complications and undergoing laparotomy or orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 50 years old
* ASA (American Society of Anaesthesiologists) Physical Status III
* Patient with increased risk of perioperative cardiac complications (Revised Cardiac Risk Index>=2)
* Surgical operation: laparotomy or orthopaedic surgery or laparoscopy
* Planned duration of general anaesthesia in the range of 2-6 hours
* Patient willing and able to complete the requirements of this study including the signature of the written informed consent

Exclusion Criteria:

* Patient with severe impairment of cardiac function (Left Ventricular Ejection Fraction < 35%)
* Patient with drug-eluting stent placed within 12 months prior to selection
* Woman of child-bearing potential not implementing adequate contraceptive methods
* Pregnant or lactating woman
* Surgical procedure in emergency
* Chronic opioids pain therapy
* Serious illness or medical conditions which are possible contra indication for elective general anaesthesia or administration of intra operative treatments, or which are interfering with the monitoring devices, such as:

  * Myocardial infarction within 6 months prior to selection
  * Any significant history of allergy/hypersensitivity to any drugs used during the study, to silicone or to latex
  * Severely impaired hearing
  * Known severe neurological disorders
  * Any medical condition which does not justify the trial participation in the investigator's judgement
  * General anaesthesia within 7 days prior to selection
  * Laparotomy within 3 months prior to selection, only for patients undergoing laparotomy
* History of drug abuse or psychiatric disorders which would impair the understanding of the necessary information or render medically or legally not able to give written informed consent
* Concurrent treatment with any other experimental drugs
* Participation in any other clinical trial within 4 weeks prior to selection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold BEIN, Prof Dr Med, Principal Investigator — University Hospital Schleswig-Holstein; Jens SCHOLZ, Prof. Dr Med, Study Chair — University Hospital Schleswig-Holstein
Locations (6):
- France (2):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Groupe Hospitalier Universitaire Caremeau, Nîmes
- Germany (3):
  - Evangelisches Waldkrankenhaus Berlin-Spandau, Berlin
  - BG Kliniken-Bergmannstrost, Halle
  - University Hospital Schleswig-Holstein, Kiel
- Manchester Royal Infirmary, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Xenon 50% (45%-55%) in Oxygen (45%-55%)
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 32 | 37 | 33
Completed | 31 | 32 | 32
Not Completed | 1 | 5 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was done in the Intention To Treat (ITT) Data Set (Randomised Patients).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 32 | 37 | 33 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (8.2) | 70.0 (9.7) | 71.1 (6.9) | 70.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 12 | 34
  Male | 22 | 25 | 21 | 68
Weight [Mean (Standard Deviation); unit: kg] | 81.18 (17.39) | 80.41 (19.61) | 81.12 (16.74) | 80.88 (17.85)
Height [Mean (Standard Deviation); unit: cm] | 168.4 (8.8) | 168.0 (8.9) | 169.2 (9.8) | 168.5 (9.1)
Body Surface Area [Mean (Standard Deviation); unit: m2] | 1.938 (0.228) | 1.926 (0.251) | 1.943 (0.228) | 1.935 (0.235)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m2] | 28.71 (6.26) | 28.43 (6.09) | 28.39 (5.98) | 28.51 (6.05)
Planned High-Risk Surgical Procedures [Number; unit: participants]
  No | 4 | 4 | 4 | 12
  Yes | 28 | 33 | 29 | 90
History of Ischemic Heart Disease [Number; unit: participants]
  No | 9 | 14 | 11 | 34
  Yes | 23 | 23 | 22 | 68
History of Congestive Heart Failure [Number; unit: participants]
  No | 23 | 28 | 22 | 73
  Yes | 9 | 9 | 11 | 29
History of Cerebrovascular Disease [Number; unit: participants]
  No | 27 | 27 | 21 | 75
  Yes | 5 | 10 | 12 | 27
Pre-Operative Treatment With Insulin or Antidiabetics [Number; unit: participants]
  No | 20 | 24 | 25 | 69
  Yes | 12 | 13 | 8 | 33
Pre-Operative Serum Creatinine >2.0 mg/dL [Number; unit: participants]
  No | 29 | 33 | 28 | 90
  Yes | 3 | 4 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Dose of Propofol (mg) Administered During Maintenance Adjusted to Patient Body Surface Area (BSA in m²) and Maintenance Duration (Min)
Description: Dose of propofol administered with a Target Controlled Infusion (TCI) device, cerebral concentration equal to 5 µg/mL at the end of induction, and then concentration adjusted to the level of depth of anaesthesia during maintenance. Depth of anaesthesia continuously assessed by signals derived from electroencephalographic recording. Analgesia during induction and maintenance obtained with remifentanil administered with a second TCI device at the stable cerebral concentration of 7 ng/mL.
Time Frame: Maintenance period (1 Day)
Population: The main analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: mg adjusted
Groups:
- Group B: Xenon 70%(65%-75%) in Oxygen (25%-35%)
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 29 | 33 | 30
mg adjusted | 1.683 (0.834) | 1.005 (1.121) | 3.987 (1.431)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; The dose of propofol adjusted to BSA and maintenance duration was expected to be 4.0 mg/m².min in the control group, 2.8 mg/m².min in one xenon group and 3.0 mg/m².min in the other xenon group. With an expected common standard deviation of 2.0 mg/m².min, a type I error of 0.05 (two-sided) and a power of 0.80, the sample size required to show a statistically significant difference between the three groups was estimated to be 48 patients per group, resulting in a total of 144 randomised patients; Test type: Superiority or Other; p < 0.0001, ANCOVA; The analysis of covariance was adjusted for quantity of propofol (mg) administered during the induction period, gender, type of surgery and centre
Statistical Analysis 2: Comparison: Group B vs Group C; Test type: Superiority or Other; p < 0.0001, ANCOVA — Pairwise comparison performed using Tukey's test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.0256, 95% CI 2-sided [2.328 to 3.724] — The difference Xenon 70% in Oxygen minus Medical Air in Oxygen was assessed
Statistical Analysis 3: Comparison: Group A vs Group C; Test type: Superiority or Other; p < 0.0001, ANCOVA — Pairwise comparison performed using Tukey's test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.2905, 95% CI 2-sided [1.570 to 3.011] — The difference Xenon 50% in Oxygen minus Medical Air in Oxygen was assessed
Statistical Analysis 4: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 0.0365, ANCOVA — Pairwise comparison was performed using the Tukey's test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.7351, 95% CI 2-sided [0.038 to 1.432] — The difference Xenon 70% in Oxygen minus Xenon 50% in Oxygen was assessed

2. Secondary Outcome: Anaesthesia Recovery Time
Description: Time interval between the end of maintenance period and time of tracheal tube removal.
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 32 | 35 | 32
minutes | 9.3 (15.8) | 22.2 (62.6) | 43.3 (180.6)

3. Secondary Outcome: Awakening Time
Description: Time interval between the end of maintenance period and time of Aldrete score ≥ 9.
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 26 | 27 | 27
minutes | 53.9 (37.6) | 70.7 (74.2) | 62.6 (34.3)

4. Secondary Outcome: Stay in the Operating Room
Description: Time interval between admission in the operating room and discharge from the operating room.
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 32 | 37 | 33
minutes | 273.1 (115.5) | 288.2 (119.1) | 315.0 (141.5)

5. Secondary Outcome: Stay in the Recovery Room
Description: Time interval between admission in the recovery room and discharge from the recovery room.
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 28 | 34 | 29
minutes | 187.5 (156.3) | 180.7 (132.0) | 218.0 (243.7)

6. Secondary Outcome: Haematology - Leucocytes (Giga/L)
Description: Leucocytes (Giga/L) obtained from blood samples collected at baseline and in the morning following surgery.
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: Giga/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 28 | 32 | 28
Giga/L
  Before Anaesthesia | 8.118 (2.289) | 8.301 (2.980) | 7.432 (1.641)
  Morning Following Surgery | 11.429 (2.737) | 11.574 (4.438) | 11.280 (2.818)

7. Secondary Outcome: Haematology - Erythrocytes (Tera/L)
Description: Erythrocytes (Tera/L) obtained from blood samples collected at baseline and in the morning following surgery.
Time Frame: 1 Postoperative Day.
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: Tera/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 28 | 32 | 28
Tera/L
  Before Anaesthesia | 4.373 (0.553) | 4.219 (0.798) | 4.135 (0.450)
  Morning Following Surgery | 3.690 (0.529) | 3.763 (0.524) | 3.675 (0.564)

8. Secondary Outcome: Haematology - Platelets (Giga/L)
Description: Platelets (Giga/L) obtained from blood samples collected at baseline and in the morning following surgery
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: Giga/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 28 | 32 | 28
Giga/L
  Before Anaesthesia | 225.036 (89.556) | 244.656 (71.724) | 244.214 (80.484)
  Morning Following Surgery | 188.036 (79.083) | 212.594 (79.424) | 196.250 (86.871)

9. Secondary Outcome: Serum Chemistry - AST (GOT) (IU/L)
Description: AST (GOT) (IU/L) obtained from blood samples collected at baseline and in Morning following surgery.
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 24 | 28 | 26
IU/L
  Before Anaesthesia | 28.641 (32.661) | 31.926 (25.495) | 30.544 (27.369)
  Morning Following Surgery | 44.723 (66.482) | 139.163 (420.704) | 62.348 (65.231)

10. Secondary Outcome: Serum Chemistry - ALT (GPT) (IU/L)
Description: ALT (GPT) (IU/L) obtained from blood samples collected at baseline and in Morning following surgery
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 23 | 28 | 28
IU/L
  Before Anaesthesia | 28.498 (31.981) | 24.400 (13.176) | 28.655 (27.587)
  Morning Following Surgery | 50.634 (111.748) | 81.747 (197.209) | 48.115 (57.414)

11. Secondary Outcome: Serum Chemistry - Gamma GT (IU/L)
Description: Gamma GT (IU/L) obtained from blood samples collected at baseline and in Morning following surgery
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 23 | 27 | 26
IU/L
  Before Anaesthesia | 122.689 (335.374) | 77.012 (80.051) | 136.785 (370.826)
  Morning Following Surgery | 106.234 (198.074) | 73.021 (86.695) | 90.345 (189.828)

12. Secondary Outcome: Serum Chemistry - Creatinine (Mcmol/L)
Description: Creatinine (mcmol/L) obtained from blood samples collected at baseline and in Morning following surgery
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 28 | 32 | 28
mcmol/L
  Before Anaesthesia | 94.625 (66.513) | 106.825 (68.814) | 98.830 (40.639)
  Morning Following Surgery | 115.007 (144.682) | 102.071 (61.185) | 96.273 (38.996)

13. Secondary Outcome: Serum Chemistry - Urea (mmol/L)
Description: Urea (mmol/L) obtained from blood samples collected at baseline and in Morning following surgery
Time Frame: 1 Postoperative Day
Population: The analysis was done in the ITT Data Set (Randomised Patients).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 24 | 27 | 22
mmol/L
  Before Anaesthesia | 7.453 (4.623) | 8.680 (5.882) | 7.886 (3.087)
  Morning Following Surgery | 7.317 (5.458) | 7.964 (4.404) | 7.609 (2.876)

ADVERSE EVENTS:
Time Frame: Adverse Events observed between the onset of induction and the study end
Description: Participants at risk are the patients from the ITT Data Set (Randomised Patients).
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 4/32 | 7/37 | 5/33
Other Adverse Events (participants affected / at risk) | 31/32 | 30/37 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=32) | Group B (N=37) | Group C (N=33)
Abdominal Sepsis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound Decomposition (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oxygen Saturation Decreased (Investigations) | 0 | 1 | 0
PO2 Decreased (Investigations) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 1
Death (General disorders) | 0 | 1 | 0
Multi-organ Failure (General disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Gastrointestinal Necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 0 | 1
Hepatobiliary Disorders (Hepatobiliary disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=32) | Group B (N=37) | Group C (N=33)
Hypotension (Vascular disorders) | 22 | 20 | 20
Hypertension (Vascular disorders) | 9 | 7 | 9
Nausea (Gastrointestinal disorders) | 7 | 9 | 5
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3
Constipation (Gastrointestinal disorders) | 3 | 2 | 4
Procedural Hypotension (Injury, poisoning and procedural complications) | 3 | 7 | 4
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 5 | 3
Anaesthetic Complication Cardiac (Injury, poisoning and procedural complications) | 1 | 3 | 0 — corresponds to 1 event of "intraoperative bradycardia"
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 2 | 1 — Corresponds to 1 event of "CK rise post-operatively" (Xenon 70%group), 1 event of "slow to breathe deeply post-operatively" (Xenon 70% group) and 1 event of "post-operative bradycardia" (Medical Air group)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 | 2 | 2
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 2
Myoglobin Blood Increased (Investigations) | 3 | 6 | 5
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 3 | 4
White Blood Cell Count Increased (Investigations) | 1 | 2 | 1
Aspartate Aminotransferase Increased (Investigations) | 2 | 1 | 2
Gamma-glutamyltransferase Increased (Investigations) | 1 | 0 | 2
Haematocrit Decreased (Investigations) | 1 | 0 | 2
Platelet Count Decreased (Investigations) | 1 | 0 | 2
Troponin T Increased (Investigations) | 1 | 0 | 2
Pain (General disorders) | 5 | 5 | 7
Hypothermia (General disorders) | 2 | 2 | 3
Hyperthermia (General disorders) | 2 | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 6 | 4 | 6
Leukocytosis (Blood and lymphatic system disorders) | 4 | 2 | 2
Bradycardia (Cardiac disorders) | 2 | 2 | 3
Tachycardia (Cardiac disorders) | 1 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Confusional State (Psychiatric disorders) | 2 | 1 | 4
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1

LIMITATIONS AND CAVEATS:
The study has been terminated earlier due to difficulties to find patients meeting the inclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days